CLINICAL TRIAL: NCT00493727
Title: Use of Mucomyst (NAC) to Ameliorate Oxidant Stress in Diabetic Patients as Measurable by Surrogate Serum Markers
Brief Title: Use of Mucomyst to Ameliorate Oxidant Stress in Diabetics With Proteinuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: West Virginia University (Other)
Responsible Party: Saklayen, Mohammad - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0030
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes; Proteinuria
Keywords: Oxidative stress; N-acetylcysteine; NAC; Isoprostane; Proteinuria; Diabetes; Mucomyst; albuminuria
MeSH Terms: conditions — Diabetes Mellitus; Proteinuria; Albuminuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: N-acetylcysteine(Mucomyst)

INTERVENTIONS:
Drug: N-acetylcysteine(Mucomyst)

SUMMARY:
The study will look at the effect of 30 days of treatment of 15 diabetics with proteinuria with N-acetylcysteine ( Mucomyst ) at a dose of 1 gm twice a day by mouth. The primary outcome that will be measured is change in the oxidant stress as measurable by changes in the serum level of isoprostane, Glutathione peroxidase, aconitase and Total oxidant stress. Secondary outcomes measured will be changes in proteinuria and kidney function as measured by spot urine pr/cr and estimated GFR by MDRD formula.

DETAILED DESCRIPTION:
Mucomyst (Acetylcysteine) for amelioration of diabetic nephropathy

Hypothesis:

Treatment with Mucomyst over several months will reduce the oxidant stress and thereby reduce the proteinuria and the progression of renal failure in patients with diabetic nephropathy.

Rationale:

Mucomyst or Acetylcysteine has now been found to be beneficial in ameliorating radio-contrast induced acute renal failure in several different studies (ref 1) The beneficial effects of Mucomyst is most likely due to its antioxidative properties. Oxidative stress plays a major role in diabetic complication especially in diabetic nephropathy.

In a recent in vitro study Acetylcysteine ameliorated the deleterious effects of albumin on cultured renal proximal tubular epithelial cells. Murine proximal tubular cells were treated with albumin (30 mg/ml medium) for various lengths of time. The results showed that albumin could activate Stat1 and Stat5 within 15 min in proximal tubular cells. The activation of STATs was mediated mostly by Jak2 and required no protein synthesis. In addition, activation of Stat1 occurred even after neutralization of IFN- . The activation of STATs was inhibited by N-acetyl-L-cysteine, a precursor of glutathione and a reactive oxygen species (ROS) scavenger, and fluorescence-activated cell sorter analysis showed upregulation of intracellular ROS after albumin overloading, suggesting that albumin per se could generate ROS in proximal tubular cells. The activation of STATs occurred by way of the ROS generating system, and especially through the membrane-bound NADPH oxidase system. Reduced activities of glutathione peroxidase and catalase could also be responsible for the accumulation of intracellular ROS. Hence, not only the ROS generating system, but also the ROS scavenging system may contribute to the induction of ROS by albumin.

N-acetylcysteine also may attenuate the course of hepatorenal syndrome, a renal vasoconstrictive response of indeterminate nature that develops during advanced liver failure. This effect, shown in experimental settings [9] and in a preliminary clinical report [10], could imply a better preservation of liver function. However, direct renal protective mechanisms may play a role also, considering the ubiquitous distribution of acylases that catalyze the deacetylation of NAC [11]. Indeed, recent studies suggest that NAC may increase intracellular glutathione and ameliorate renal ischemia-reflow injury [12-14], inferior vena cava-occlusion [15] or kidney damage from cis-platinum [16], cyclosporine [17], and other nephrotoxic insults [18, 19]. NAC has been reported recently to prevent radiocontrast nephropathy in high-risk patients [20]. These studies, conducted in a clinical trial without preliminary experiments in animals, underscore the safety of oral NAC administration.

As stated above, the mechanism of NAC-related organ protection is primarily attributed to scavenging oxygen free radicals, either directly, or through increasing intracellular glutathione concentration [3, 4]. Indeed, decreased malonaldehyde production indicates an attenuation of membrane damage from oxygen-free radicals [3], but other protective mechanisms may play a role as well [21]. Improved local microcirculation may be a major potential NAC-related organ-protective mechanism. NAC was reported to augment papillary flow [22] and was found to improve renal vasodilation in response to acetylcholine [15]. Thus, perhaps some of the protective effects of NAC can be attributed to improved glomerular hemodynamics or to the prevention of hypoxic tubular damage via restoration of altered renal microcirculation.

NAC ameliorates renal vasoconstriction, an effect that seems to be mediated by mechanisms other than prostaglandins and nitric oxide

NAC had been safely used in a large group of ESRD patients for over one year ( 600 mg bid by mouth ) in a prospective randomized trial . The group treated with NAC had reduction in composite cardiovascular endpoints ( 18% vs 47%) ( Ref: Circulation2003,107: 992 . Tepel et al )

Similarly in a RCt of Alzheimer patients NAC treatment for 6 months showed benefit in cognitive tasks in the treatment group. ( Ref: Neurology2001, 23: 57: Adair et al )

Intravenous injection of NAC prior to dialysis increased the dialysis clearance of homocysteine and improved endothelial function in a group of ESRD patient ( Ref: Circulation 2003, 109: 369; Scholze et al )

NAC treatment was also found to have potentiating effect of the antihypertensive effects of ACE inhibitors in hypertensive patients ( Blood pressure 2002, 11:235; Barrios et al )

In another RCT in an aging population, chronic treatment with NAC was seen to cause significant decrease in plasma TNF-alpha and improved the muscle strength. ( Ref: J Mol MED 2003; 81: 118; Hauer et al.)

Protocol:

All patients with diabetes and proteinuria at any level will be eligible for the study. Patients who are on dialysis and who have known allergy to Mucomyst will be excluded

Patients will get Mucomyst 1000 mg by mouth twice a day for 30 days. Urine and serum will be collected at the beginning, , at 15 and 30 days after starting Mucomyst and 30 days after stopping Mucomyst. Portions of the blood and urine will be frozen and mailed to a special lab to measure the chemicals that determine the level of oxidative stress. The particular chemicals that will be tested for are isoprostane in urine and isoprostane, aconitase, glutathione peroxidase and total serum antioxidant stress in the blood. The special tests will be done by Dr. Valyathan's lab . Locally we will test blood and urine for proteinuria and kidney Fx.

.

Data collection:

Demographic information:

Wt, BP at every visit:

Med list rechecked at every visit:

At every visit:

Collection of blood for different measures of oxidant stress: serum will be frozen to be sent to Dr. Vallyathan's lab later.

Blood for renal function test

Spot urine protein/cr (quantitative proteinuria) and also for measuring isoprostane

Outcome:

The primary outcome will be the reduction in the measured oxidant stress markers in the serum such as isoprostane, glutathione peroxidase, aconitase, and total oxidant stress. Secondary outcome will be reduction in proteinuria and the change in kidney function during treatment with Mucomyst.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic with proteinuria

Exclusion Criteria:

* Allergy to mucomyst and pt on dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
This research will test the possibility the Mucomyst given by mouth for a month will decrease oxidative stress and slow the disease.

SECONDARY OUTCOMES:
Reduction of proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad G. Saklayen, MD, Principal Investigator — VA Medical Center, Dayton
Locations (1):
- VA Medical Center, Dayton, Dayton, Ohio, United States